CLINICAL TRIAL: NCT07029607
Title: A Randomized Double Blind, Placebo Controlled Clinical Study Evaluating the Efficacy and Safety of Magnesium Supplementation on Relaxation in Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olly, PBC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OLLCLI2F
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Healthy
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Oral dietary supplement. Instructions: Take 4 gummy per day with or without food or water. Chew thoroughly before swallowing. Do not take more than 4 gummy per day.
  Interventions: Dietary Supplement: Placebo
- Dietary Supplement with actives (Active Comparator): Oral dietary supplement. Instructions: Take 4 gummy per day with or without food or water. Chew thoroughly before swallowing. Do not take more than 4 gummy per day.
  Interventions: Dietary Supplement: Dietary Supplement with actives

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo
  Arms: Placebo
Dietary Supplement: Dietary Supplement with actives — Dietary Supplement containing magnesium
  Arms: Dietary Supplement with actives

SUMMARY:
The study will assess the efficacy of magnesium supplementation for improvement of body and mind relaxation (through stress levels), and sleep score compared to placebo, assessed by validated questionnaires. Participants will be asked to take the supplement every day for 12 weeks and will complete monthly check-ins and questionnaires. Participants will monitor adverse events in a journal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants (women + men)
* Will maintain regular diet and exercise habits
* Agreement to adhere to the procedures and requirements of the study and to report to the institute on the day(s) and at the time(s) scheduled for the assessments.

Exclusion Criteria:

1. Neurological or psychiatric disorders
2. Pregnant or breastfeeding
3. Known allergies to magnesium-containing products
4. Taking a medication known to interact with magnesium, or taking loop diuretics, cyclosporine, digoxin, amphotericin.
5. No concurrent magnesium supplementation
6. Substance or alcohol abuse
7. Currently use, or have used within appropriate washout period, any prescription, over the counter medication, or supplements with primary CNS activity such as Antidepressants,mood stabilizer and anxiolytics, Sedatives and Stimulants
8. Anticholinergic or cholinergic medications
9. Anti-inflammatory and analgesic medication (except for PRN use)
10. Anti-allergy medication (except for non-sedating antihistamines)
11. Blood thinners
12. Other prescribed medications that may affect cognition, stress, or mood
13. Body mass index (BMI) greater than 40 kg/m2 ,
14. Individuals on angiotensin converting enzyme inhibitors for blood pressure control, other magnesium-retaining drugs, or potassium-sparing drugs
15. History of reaction to the category of product tested
16. Other diseases or medications that might directly interfere in the study or put the subject's health under risk.
17. Subjects with any invasive medical procedures during the study.
18. Participants who are unreliable or unlikely to be available for the duration of the study.
19. No employees of PCR or the sponsor (e.g OLLY PBC, Unilever, or the H&W Collective)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-14 (Estimated); Primary Completion 2025-10-06 (Estimated); Study Completion 2025-10-24 (Estimated)

PRIMARY OUTCOMES:
Changes in PSS scores | From start of study until end of the study at week 12
  Monthly PSS scores will be analyzed to assess changes in stress levels across the actives and the placebo

SECONDARY OUTCOMES:
Changes in Relaxation State Questionnaire scores | From start of study until end of the study at week 12
  Monthly RSQ scores will be analyzed to assess the changes in mind and body relaxation levels across the actives and placebo

OTHER OUTCOMES:
Changes in PSQI levels | From start of study until end of the study at week 12
  Monthly PSQI scores will be analyzed to assess the changes sleep quality across the actives and placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Princeton Consumer Research, St. Petersburg, Florida, United States